CLINICAL TRIAL: NCT01569841
Title: A Trial Comparing the Efficacy of Insulin Degludec With Insulin Glargine on Glycaemic Control Using Continuous Glucose Monitoring in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3874; U1111-1125-7495 (Other: WHO)
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg (Experimental)
  Interventions: Drug: insulin degludec
- IGlar (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Administered subcutaneously (s.c., under the skin) once daily.
  Arms: IDeg
Drug: insulin glargine — Administered subcutaneously (s.c., under the skin) once daily.
  Arms: IGlar

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to compare the efficacy of insulin decludec with insulin glargine on glycaemic control using continuous glucose monitoring in patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* HbA1c (glycosylated haemoglobin) below or equal to 8.5%
* Current treatment with IGlar (insulin glargine) in a basal-bolus regimen with a total daily dose below 120 U
* BMI (body mass index) below 35 kg/m^2

Exclusion Criteria:

* Use within the last 3 months prior to visit 1 (screening) of any antidiabetic glucose lowering drug other than insulin/insulin analogues
* Subjects with regular use of acetaminophen who are not willing to use another analgetic during CGM (Continuous Glucose Monitoring) periods
* Stroke; heart failure; myocardial infarction; unstable angina pectoris; coronary arterial bypass graft or angioplasty within 24 weeks prior to visit 1
* Recurrent severe hypoglycemia (more than one severe hypoglycemic event during the last 12 months) or hypoglycemia unawareness or hospitalization for diabetic ketoacidosis during the previous 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Clinical Trial Call Center, Minneapolis, Minnesota, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at one site in the United States of America (USA).
Pre-assignment Details: All subjects were on basal-bolus insulin regimens at screening using insulin glargine (IGlar) and either insulin aspart (IAsp) or insulin lispro (ILis). During the run-in period, IGlar 100 U/mL was administered subcutaneously (under the skin) once daily (OD) in the morning (before breakfast) along with IAsp 100 U/mL as meal-time insulin.
Groups:
- IDeg/IGlar: The trial included 2 treatment periods of 6 weeks each in a cross-over design, and a follow-up visit no less than 7 days after the last treatment visit. Total trial duration for the individual subject was 18 weeks.
  All randomised subjects were scheduled for 12 weeks of treatment with the trial products. After 6 weeks of treatment in period A, the subjects were crossed over to 6 weeks of the other treatment in period B.
  Upon completing the 4-week run-in period, subjects randomised to the IDeg/IGlar treatment sequence received an morning dose of IDeg OD (100 U/mL, 3 mL prefilled pen) along with mealtime dosing of IAsp (100 U/mL, prefilled pen) subcutaneously (under the skin) for 6 weeks in treatment period A. Upon completion of treatment Period A, subjects crossed over to Period B and received a morning dose of IGlar OD (100 U/mL, SoloStar® prefilled pen) in combination with mealtime dosing of IAsp (100 U/mL, prefilled pen) subcutaneously (under the skin) for 6 weeks.
- IGlar/IDeg: The trial included 2 treatment periods of 6 weeks each in a cross-over design, and a follow-up visit no less than 7 days after the last treatment visit. Total trial duration for the individual subject was 18 weeks.
  All randomised subjects were scheduled for 12 weeks of treatment with the trial products. After 6 weeks of treatment in period A, the subjects were crossed over to 6 weeks of the other treatment in period B.
  Upon completing the 4-week run-in period, subjects randomised to the IGlar/IDeg treatment sequence received an morning dose of IGlar OD (100 U/mL, 3 mL SoloStar® prefilled pen) subcutaneously (under the skin) in combination with mealtime dosing of IAsp (100 U/mL, prefilled pen) for 6 weeks in treatment Period A. Upon completion of treatment Period A, subjects crossed over to Period B and received a morning dose of IDeg OD (100 U/mL, 3 mL prefilled pen) subcutaneously (under the skin) in combination with mealtime dosing of IAsp (100 U/mL, prefilled pen) for 6 weeks.
Period: Period A (6 Weeks)
Arm/Group | IDeg/IGlar | IGlar/IDeg
Started | 12 | 12
Exposed | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period B (6 Weeks)
Arm/Group | IDeg/IGlar | IGlar/IDeg
Started | 12 | 11
Exposed | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Full Analysis Set: The full analysis set (FAS) included all randomised subjects.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 10.7 (3.4)
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.1 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Average Time Within Glycaemic Target Range (Above 70 mg/dL and Below 130 mg/dL)
Description: Time within the glycaemic target range [> 70 mg/dL (3.9 mmol/L) and < 130 mg/dL (7.2 mmol/L)] measured by Continuous Glucose Monitoring (CGM) in the last four hours of each dosing interval during the last 2 weeks of the 6-week treatment period.
Time Frame: CGM occured during the last 2 weeks of the 6 weeks treatment period.
Population: The FAS included all randomised subjects. One subject from the IGlar to IDeg treatment sequence withdrew from the trial during treatment period A while taking IGlar.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- IDeg: The trial included a screening period of approximately one week, a run-in period of 4 weeks followed by 2 treatment periods of 6 weeks each in a cross-over design, and a follow-up visit no less than 7 days after the last treatment visit. Total trial duration for the individual subject was 18 weeks.
  Treatment period A: Subjects from run-in period were randomised to insulin degludec (IDeg) OD (100 U/mL, 3 mL prefilled pen, morning dose) administered subcutaneously (under the skin) in combination with mealtime IAsp (100 U/mL, pre-filled pen) for 6 weeks.
  Treatment period B: Subjects (from treatment period A) were crossed over to IGlar OD (100 U/mL, SoloStar® prefilled pen, morning dose) in combination with mealtime IAsp (100 U/mL, s.c., prefilled pen) for 6 weeks.
- IGlar: The trial included a screening period of approximately one week, a run-in period of 4 weeks followed by 2 treatment periods of 6 weeks each in a cross-over design, and a follow-up visit no less than 7 days after the last treatment visit. Total trial duration for the individual subject was 18 weeks.
  Treatment period A: Subjects from run-in period were randomised to IGlar OD (100 U/mL, 3 mL SoloStar® prefilled pen s.c., morning dose) in combination with mealtime IAsp (100 U/mL, prefilled pen s.c.) for 6 weeks.
  Treatment period B: Subjects (from treatment period A) were crossed over to IDeg OD (100 U/mL, prefilled pen s.c., morning dose) for 6 weeks in combination with mealtime IAsp (100 U/mL, prefilled pen s.c.) for 6 weeks.
Arm/Group | IDeg | IGlar
Number analyzed (Participants) | 23 | 23
hours | 1.39 (0.71) | 1.09 (0.77)

2. Secondary Outcome: Mean Interstitial Glucose (IG) Based on 14 Days of CGM
Description: The observed mean of IG profile was obtained as the average value of area under the IG profile divided by the actual assessment time interval during the last 2 weeks of the 6-week treatment period.
Time Frame: CGM monitoring occurred during the last 2 weeks of the 6-week treatment period.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg | IGlar
Number analyzed (Participants) | 23 | 23
mmol/L | 9.6 (1.5) | 9.8 (1.7)

3. Secondary Outcome: Fasting Plasma Glucose (FPG)
Description: FPG after 6 weeks of treatment in each treatment period.
Time Frame: At the end of each 6 week treatment period.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg/IGlar | IGlar/IDeg
Number analyzed (Participants) | 12 | 11
mmol/L
  Treatment period A | 8.8 (4.6) | 10.9 (4.8)
  Treatment period B | 10.4 (3.4) | 10.9 (4.4)

4. Secondary Outcome: Glycosylated Haemoglobin (HbA1c)
Description: HbA1c after 6 weeks of treatment in each treatment period.
Time Frame: At the end of each 6 week treatment period.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg/IGlar | IGlar/IDeg
Number analyzed (Participants) | 12 | 11
percentage of glycosylated haemoglobin
  Treatment period A | 6.6 (0.5) | 7.1 (0.6)
  Treatment period B | 6.9 (0.7) | 7.3 (0.6)

5. Secondary Outcome: Number of Treatment Emergent Adverse Events (AEs)
Description: Number of treatment emergent adverse events (TEAEs). An AE was defined as treatment emergent if the onset date was on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment. Severity was assessed by investigator.
Time Frame: Within each week 6 treatment period
Population: The safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: events
Arm/Group | IDeg | IGlar
Number analyzed (Participants) | 23 | 24
events
  Adverse Events | 18 | 16
  Serious Adverse Events | 0 | 0
  Severe Adverse Events | 3 | 0
  Moderate Adverse Events | 5 | 0
  Mild Adverse Events | 10 | 16
  Fatal Adverse Events | 0 | 0

6. Secondary Outcome: Number of Treatment Emergent Confirmed Hypoglycaemic Episodes
Description: A hypoglycaemic episode was defined as treatment emergent if the onset of the episode occurred after the first administration of investigational medicinal product (IMP), and no later than 7 days after the last day on trial product. Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia or minor hypoglycaemic episodes. Severe hypoglycaemic episodes: requiring assistance to administer carbohydrate, glucagon or other resuscitative actions. Minor hypoglycaemic episodes: able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Hypoglycemic episodes reported within each 6 week treatment period.
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: events
Arm/Group | IDeg | IGlar
Number analyzed (Participants) | 23 | 24
events | 283 | 239

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected during each 6 week treatment period + 7 days follow up.
Description: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg | IGlar
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 8/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg (N=23) | IGlar (N=24)
Nasopharyngitis (Infections and infestations) | 0 (0) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of plans by any investigator to publish and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to Novo Nordisk before submission for comments. Comments will be given within four weeks from receipt of the planned communication.